CLINICAL TRIAL: NCT05165030
Title: Identification of Genetic Mutations Involved in Chiari Type I Malformations
Acronym: ChiariGene
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP210472
Record Dates: First submitted 2021-10-28; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-10

CONDITIONS: Chiari Malformation, Type 1
Keywords: genetic mutation; syringomyelia
MeSH Terms: conditions — Arnold-Chiari Malformation; Syringomyelia | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Blood sample for all participant during a consultation specific for the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood Sample (Experimental): Blood Sample
  Interventions: Genetic: Blood Sample

INTERVENTIONS:
Genetic: Blood Sample — clinical-radiological evaluation, genetic analysis by whole exome sequencing and constitution of a bio-collection

SUMMARY:
Although most cases of Chiari malformation type I (CM1) are sporadic, familial cases of CM1, with or without syringomyelia, suggest a genetic cause in the pathogenesis of these malformations.

The hypothesis is that there is one or more genes, in particular among those involved in the development of the axial skeleton and the cranium, which could lead to an abnormal morphology of the posterior fossa resulting in tonsillar herniation defining CM1.

The abnormal circulation of cerebrospinal fluid due to tonsillar herniation is believed to be responsible, in some patients whose predisposing factors remain to be determined, for the progressive onset of associated syringomyelia.

Since the determinants underlying the development of the posterior fossa of the skull are multigenic, the analysis of familial cases would make it possible to reduce genetic and phenotypic heterogeneity allowing to identify common pathogenic variants.

For this study the investigators will be taking a blood sample to perform whole exome sequencing, build a biological collection and record imaging and clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Having a social security
* Participant or legal representative having given his consent
* For patients: Diagnosis of a Chiari malformation type 1, defined morphologically as cerebellar tonsillar herniation beyond the foramen magnum greater than 5 mm, with or without associated syringomyelia, and which has at least one relating to the 1st or 2nd degree (parents, siblings; grandparents, uncles, aunts, cousins) carrying the malformation.
* For relatives: at least two 1st degree relatives diagnosed with a Chiari type 1 malformation

Exclusion Criteria:

* Syndromic form of Chiari malformation
* Patient with a legal protection measure
* Pregnant or breastfeeding woman
* Contraindication to MRI
* For patients: diagnosis of Chiari malformation type 1 that could not be confirmed by MRI
* For relatives: age under 18 years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Identification of the gene (s) whose mutations are responsible for the occurrence of a Chiari type I malformation, whether associated with syringomyelia or not. | At inclusion (as soon as the patient agree)
  Description of gene mutations in patients with Chiari type I malformation by whole exome sequencing

SECONDARY OUTCOMES:
Identification of the gene (s) whose mutations are associated with the occurrence of syringomyelia in patients with Chiari type I malformation | At inclusion (as soon as the patient agree)
  Description of gene mutations in patients with syringomyelia associated with Chiari type I malformation
Establishment of a DNA bank for familial Chiari type I malformations | At inclusion (as soon as the patient agree)
  Bio-collection

CONTACTS AND LOCATIONS:
Overall Officials: Steven Knafo, Principal Investigator — APHP
Locations (1):
- Service de Neurochirurgie, Le Kremlin-Bicêtre, Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No